CLINICAL TRIAL: NCT05707143
Title: Comparative Effects of Home Based Stabilization and Kegel Exercises on Low Back Pain, Disability and Quality of Life in Postnatal Females
Brief Title: Effects of Home Based Stabilization and Kegel Exercises on Postnatal Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mehak Hassan
Record Dates: First submitted 2023-01-23; First posted 2023-01-31 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: disability; low back pain; females; quality of life; stabilization exercises
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- home based stabilization exercises (Active Comparator): knee rolls, the cat, spine curl, bridging, single knee to chest, pelvic tilt
  Interventions: Other: home based stabilization exercises
- kegel exercises (Experimental): kegel exercises
  Interventions: Other: kegel exercises

INTERVENTIONS:
Other: home based stabilization exercises — 3 times per day with 10 repetitions and holding time will be 5-10 sec
  Arms: home based stabilization exercises
Other: kegel exercises — 3 times per day with 10 repetitions and holding time will be 5-10 sec
  Arms: kegel exercises

SUMMARY:
To compare the effects of home based stabilization exercises and kegel exercises on low back pain, disability and quality of life in postnatal females.

ELIGIBILITY:
Inclusion Criteria:

* Cesarean delivery.
* Multi gravida females.
* Postpartum low back pain last for 1 year

Exclusion Criteria:

* Low back pain before pregnancy.
* Urogenital infections.
* History of pelvic floor or lumber surgery.
* Malignancy.
* Pelvic or lumber fractures

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — post partum females
Enrollment: 22 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale | 6th week
  A tool used to help a person rate the intensity of pain. The visual analogue scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. High reliability when it is used for acute abdominal pain and moderate to good reliability for disability in patient with chronic musculoskeletal pain. It is a validated, subjective measure for acute and chronic pain
Short form 36 | 6th week
  The Short form 36 health survey questionnaire is used to indicate the health status of particular population, to help with service planning and to measure the impact of clinical and social intervention.
  The SF-36 is considered to be a valid, reliable, concise and generic measure of state of health
Oswestry disability index | 6th week
  The Oswestry disability index is a self-rating condition-specific outcome measure for evaluation of low back pain disability. It is a validated, 10-point patient-reported outcome questionnaire. It is considered the Gold standard for measuring disability and quality of life, impairment for adult with low back pain. The ODI ca be used to assess both chronic and acute conditions of varying severity. It has a high test-retest reliability and takes around 5 min for a patient to complete

CONTACTS AND LOCATIONS:
Overall Officials: Hina Gul, MS-OMPT, Principal Investigator — Riphah International University
Locations (1):
- gynecological department of Services hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khorasani F, Ghaderi F, Bastani P, Sarbakhsh P, Berghmans B. The Effects of home-based stabilization exercises focusing on the pelvic floor on postnatal stress urinary incontinence and low back pain: a randomized controlled trial. Int Urogynecol J. 2020 Nov;31(11):2301-2307. doi: 10.1007/s00192-020-04284-7. Epub 2020 Apr 10. PMID 32274521
- [Background] Urme NA, Alam F, Jahan N. Effectiveness of Specific Lumbar Stabilization Exercise for LBP among Postpartum Women: A Quasi-Experimental Study. Journal of Advanced Academic Research. 2021;8(1):79-95
- [Background] Teymuri Z, Hosseinifar M, Sirousi M. The Effect of Stabilization Exercises on Pain, Disability, and Pelvic Floor Muscle Function in Postpartum Lumbopelvic Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Dec;97(12):885-891. doi: 10.1097/PHM.0000000000000993. PMID 29979205
- [Background] Unsgaard-Tondel M, Vasseljen O, Woodhouse A, Morkved S. Exercises for Women with Persistent Pelvic and Low Back Pain after Pregnancy. Glob J Health Sci. 2016 Sep 1;8(9):54311. doi: 10.5539/gjhs.v8n9p107. PMID 27157173
- [Background] Tseng PC, Puthussery S, Pappas Y, Gau ML. A systematic review of randomised controlled trials on the effectiveness of exercise programs on Lumbo Pelvic Pain among postnatal women. BMC Pregnancy Childbirth. 2015 Nov 26;15:316. doi: 10.1186/s12884-015-0736-4. PMID 26612732